CLINICAL TRIAL: NCT07098455
Title: Comparative Effectiveness of Genicular Nerve Radiofrequency Thermocoagulation and Intra-Articular Pulsed Radiofrequency in the Management of Knee Osteoarthritis Pain
Acronym: GNRFT & IAPRF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ali ÇOŞTU, Principal investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2-25-10611
Record Dates: First submitted 2025-07-10; First posted 2025-08-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthristis; Radiofrequency Ablation
Keywords: Osteoarthritis of Knee; Pulsed Radiofrequency Treatment; Radiofrequency Ablation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNRFT - Genicular Nerve Radiofrequency Ablation (Experimental): Patients in this group will undergo ultrasound-guided genicular nerve radiofrequency ablation.
  Interventions: Procedure: GNRFT- genicular nerve radiofrequency ablation
- IAPRF - Intra-articular pulsed radiofrequency (Experimental): KNEE INTRAARTICULAR PULSED RADIOFREQUENCY WILL BE APPLIED TO PATIENTS IN THIS GROUP
  Interventions: Procedure: IAPRF- Intraarticular pulsed radiofrequency

INTERVENTIONS:
Procedure: GNRFT- genicular nerve radiofrequency ablation — Ultrasound-guided genicular nerve radiofrequency ablation will be performed
  Arms: GNRFT - Genicular Nerve Radiofrequency Ablation
Procedure: IAPRF- Intraarticular pulsed radiofrequency — Intra-articular pulsed radiofrequency will be applied under fluoroscopy guidance.
  Arms: IAPRF - Intra-articular pulsed radiofrequency

SUMMARY:
Osteoarthritis (OA) is a degenerative disease characterized by progressive cartilage deterioration, osteophyte formation, subchondral sclerosis, and a number of biochemical and morphological changes in weight-bearing joints that are affected by genetic, mechanical, and biochemical factors. The prevalence of secondary chronic knee pain in OA is more than 12% in individuals over the age of 60. It is one of the most common musculoskeletal disorders in elderly patients and has become a global health problem. Standard treatments for OA include physical therapy, nonsteroidal anti-inflammatory drugs (NSAIDs), tramadol, opioids, intra-articular hyaluronic acid, or steroids. In more severe cases, surgical knee arthroplasty should be considered. But long-term use of NSAIDs is associated with stomach bleeding, adverse cardiovascular events, and kidney failure. Opioids are often used, but a large number of side effects are encountered, especially in the elderly. Knee surgery is not always possible and can cause complications such as hematomas, infections, and damage to the surrounding tissue.

Radiofrequency (RF) application (pulsed or continuous) is a neuromodulatory or neurolytic technique that represents an alternative in pain due to osteoarthritis. RF therapy is one of the conservative treatments that has many advantages, such as minimal invasiveness, rapid recovery, and less negative response. Radiofrequency thermocoagulation (RFT) destroys the integrity of peripheral nerves using hyperthermia and thereby blocks the transmission of pain signals, while pulsed radiofrequency (PRF) regulates neurological functions or inhibits the production of immunoinflammatory factors (e.g., IL-1β, TNF-α, IL-6) by using electric fields to affect their production, thereby relieving pain in patients.

Genicular nerve radiofrequency thermocoagulation application and knee intra-articular pulsed radiofrequency application are the two radiofrequency methods routinely applied in the treatment of gonarthrosis-induced pain in our clinic. In this study, it is aimed to evaluate the effectiveness of these two methods and compare their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Patients who have pain due to knee osteoarthritis
* Patients who agree to undergo knee geniculate nerve thermocoagulation or knee intra-articular pulsed radiofrequency therapy and follow-up.

Exclusion Criteria:

* Patients using anticoagulants and those with coagulation disorders,
* Patients with psychomotor disorders,
* Patients who have undergone intra-articular injections, interventional procedures, or surgery for knee osteoarthritis in the last year,
* Patients with bacterial infection or infectious discharge in the area to be treated,
* Patients with allergies to local anesthetics, and pregnant and breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
NRS | baseline, at the 3rd month
  Pain intensity was measured using an 11-point Numeric Rating Scale, where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients rated their pain intensity based on their average pain during the defined time frame. Changes in NRS scores over time were used to evaluate treatment response.

SECONDARY OUTCOMES:
GPE | baseline, 3rd month
  Overall patient-perceived change in symptoms was assessed using the Global Perceived Effect scale. Patients rated their overall condition compared with baseline on a Likert-type scale ranging from "very much worse" to "very much improved." The GPE was used to capture the patient's global assessment of treatment effectiveness.
WOMAC | baseline; 3rd month
  Functional status was assessed using the WOMAC questionnaire, a validated disease-specific instrument for osteoarthritis. The WOMAC consists of 24 items across three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). Higher scores indicate worse pain, stiffness, and functional limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No